CLINICAL TRIAL: NCT05847244
Title: The Effect of Addition of Metformin In Obese Non- Diabetic Patients With Heart Failure With Preserved Ejection Fraction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sara ElAdawy (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Sara ElAdawy, lecturer of clinical pharmacy, October University for Modern Sciences and Arts
Organization: October University for Modern Sciences and Arts (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSPL1.5
Record Dates: First submitted 2023-04-16; First posted 2023-05-06 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Diastolic Dysfunction; Obesity
Keywords: metformin; obesity; diastolic dysfunction
MeSH Terms: conditions — Obesity | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: prospective open-label, randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): Lifestyle counseling plus standard evidence based therapy
- intervention (metformin) (Experimental): Lifestyle counseling plus standard evidence based therapy and metformin (target dose 1000 mg bid)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — The intervention will consist in giving metformin starting with 500 mg once daily (at breakfast) during the first week; if well tolerated, the dose was progressively increased to 500 mg twice daily (at breakfast and dinner) during week 2, to 1000 mg at breakfast and 500 mg at dinner during week 3, in order to reach the target dose of 1000 mg twice daily (at breakfast and dinner)
  Arms: intervention (metformin)

SUMMARY:
Diabetes mellitus people have a higher incidence of cardiovascular disease, and the results of cardiovascular events are worse. Heart failure and diabetes both have a worse prognosis, with a 1.5-2 times increased risk of death. Data from the literature have shown that MET lowers mortality by 14-35% in this patient population, which represents one-third of all HF patients with no increases in lactic acidosis incidence.

DETAILED DESCRIPTION:
Heart failure (HF) with preserved ejection fraction (HFpEF) is a distinct phenotype hallmarked by clinical signs and symptoms of HF coupled with a normal ejection faction (EF ≥ 50%) and evidence of increased left ventricular (LV) pressures and impaired LV filling on echocardiography. HFpEF is highly prevalent, accounting for up to 50% of all patients with HF, and is associated with significant morbidity and mortality. HFpEF is a heterogenous disorder, contributed to by comorbidities that include hypertension, diabetes, obesity, coronary artery disease (CAD), chronic kidney disease (CKD), and specific causes such as cardiac amyloidosis. These chronic conditions complicate the management of HF and have a significant impact on its prognosis. How to generate specific recommendations addressing many of these conditions in the setting of HF is challenging given the current state of the evidence.

Obesity is a growing global concern, and is a common finding in the progression of HFpEF. According to the World Health Organization (WHO), percentage of adult population that is obese in Egypt is 32% which makes it ranks 18th with the highest prevalence of obesity worldwide. Very few studies have been published about the burden of diseases in Egypt in general, and the burden of obesity is even more complex as the impact of obesity is a result of its comorbidities rather than a direct effect. Several studies have provided evidence for the distinct obesity related HFpEF phenotype, and its unique pathophysiology based on the obesity criteria for the European and American population with a body mass index (BMI) greater than 30 kg/m2. Obesity is a commonly occurring comorbidity in patients with HFpEF, and has many deleterious effects on the cardiovascular system, mediated by changes in volume overload, cardiac load, energy substrate utilization, tissue metabolism, and systemic inflammation. However, based on latest heart failure guidelines, evidence gaps and future research directions are needed to assess efficacy and safety of weight loss management and treatment strategies in patients with HF and obesity.

Metformin is a common anti-diabetic drug with both systemic and cardioprotective benefits in addition to its hypoglycaemic effect. At the cellular level metformin activates adenosine monophosphate-activated protein kinase (AMPK) an important regulator of several metabolic pathways resulting in enhanced glucose utilisation, reduction of protein synthesis and improvement of mitochondrial function. Furthermore, metformin has been shown to reduce collagen accumulation and potentially reduce LV hypertrophy and improve diastolic function in the diabetic myocardium. The cardio protection afforded by metformin treatment seems to result from interference with TGF-beta signaling pathway and activation of the AMP-kinase signaling cascade. A recent systematic review and meta regression analysis have shown that metformin treatment was associated with a reduction in mortality in patients with HFpEF. In addition, treatment with metformin of non-diabetic metabolic syndrome patients with diastolic dysfunction, on top of lifestyle counseling, was associated with improved diastolic function. Moreover, some studies have shown that metformin can reduce body weight. However, metformin has not been officially approved as a medicine for weight loss because its effect on different populations remains inconsistent. No studies to date assessed the role of metformin in obese non-diabetic patients with HFpEF Accordingly, investigators aimed to evaluate if metformin can improve diastolic function in non-diabetic obese patients with HFpEF. Investigators also aimed to assess the impact of this therapy in functional capacity, weight loss and health-related quality of life (HRQoL).

ELIGIBILITY:
Inclusion Criteria:

* - Inclusion criteria:

  * Age of 40 years to 74 years.
  * HFpEF (≥ 50%)
  * Written informed consent of the subject to participate in the study.
  * New York Heart Association functional class II-IV.
  * Body mass index ≥ 30 Kg/m2

Exclusion Criteria:

* - Exclusion criteria:

  * Patients with heart failure with reduced ejection fraction (< 40%)
  * Age less than 40 and more than 74
  * New York Heart Association functional class I
  * Body mass index < 30 Kg/m2
  * Diabetic patients or prior metformin user
  * Renal impairment
  * Known allergy to metformin
  * End- stage liver disease
  * Cancer
  * Pregnancy or lactation

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The change in the mean early diastolic mitral annular velocity (mean e'), at 3 and 6 months | baseline, 3 and 6 months
  Mean early diastolic mitral annular velocity assessed by echocardiography

SECONDARY OUTCOMES:
HRQOL (MLFHQ) adverse effects of metformin hospitalization rate Change in N-terminal pro-BNP (NT-proBNP) and Change in body weight | baseline, 3 and 6 months
  HRQOL using Minnesota Living with Heart Failure Questionnaire for quality-of-life evaluation (MLFHQ)
adverse effects of metformin | baseline, 3 and 6 months
  lactic acidosis side effects : dyspnea, muscle cramps, abdominal pain ,hypothermia or asthenia
hospitalization rate | baseline, 3 and 6 months
  hospitalization rate
Change in N-terminal pro-BNP (NT-proBNP) | baseline, 3 and 6 months
  Change in N-terminal pro-BNP (NT-proBNP)
Change in body weight | baseline, 3 and 6 months
  Change in body weight (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: sara Eladawy, PhD, Study Director — MSa university; Naglaa Bazan, Ass. Prof, Principal Investigator — Cairo University; shreen Elgengeehy, Prof., Study Chair — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University Hospitala, Cairo
  - Cairo University Hospitals, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pu R, Shi D, Gan T, Ren X, Ba Y, Huo Y, Bai Y, Zheng T, Cheng N. Effects of metformin in obesity treatment in different populations: a meta-analysis. Ther Adv Endocrinol Metab. 2020 May 21;11:2042018820926000. doi: 10.1177/2042018820926000. eCollection 2020. PMID 32499908
- [Result] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Result] Ladeiras-Lopes R, Sampaio F, Leite S, Santos-Ferreira D, Vilela E, Leite-Moreira A, Bettencourt N, Gama V, Braga P, Fontes-Carvalho R. Metformin in non-diabetic patients with metabolic syndrome and diastolic dysfunction: the MET-DIME randomized trial. Endocrine. 2021 Jun;72(3):699-710. doi: 10.1007/s12020-021-02687-0. Epub 2021 Apr 8. PMID 33830437
- [Result] Halabi A, Sen J, Huynh Q, Marwick TH. Metformin treatment in heart failure with preserved ejection fraction: a systematic review and meta-regression analysis. Cardiovasc Diabetol. 2020 Aug 5;19(1):124. doi: 10.1186/s12933-020-01100-w. PMID 32758236